CLINICAL TRIAL: NCT04586972
Title: Safety and Efficacy of Apixaban in Very Old Geriatric Subjects (> 80 Years) With Atrial FIbrillation in a Prospective reAl World Study;
Acronym: SOFIA
Status: Completed | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A03160-57
Record Dates: First submitted 2020-09-25; First posted 2020-10-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Nonvalvular Atrial Fibrillation
Keywords: Nonvalvular Atrial fibrillation; Apixaban.; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of this study is to realize an observational "real life" study conducted in French geriatric settings, to assess safety and efficacy in ≥ 80 year-old patients with nonvalvular Atrial fibrillation (AF) newly treated with Apixaban.

Moreover, in this geriatric population the adequacy of Apixaban dosage and events (bleeding and stroke) will be assessed.

DETAILED DESCRIPTION:
It is a muliticentric, observational, prospective study.

This study will be conducted in about 40 geriatric settings in France.

The planned duration of the inclusion period is 27 months in each center.

The follow-up period starts from inclusion up to one year after inclusion with phone contact or unscheduled visit at 3, 6, 9 and 12 months.

During this follow-up, participants physicians will record patients' data during visit directly from the patients or their physicians or their families and by phone.

The following data will be colllected:

* At M0 : Socio-demographics, clinical and biological data; embolic risk and emorrhagic risk scores,cognitive function, number of falls, blood pressure, nutritional assessment, athonomy, comorbidities, data on anticoagulant therapy, treatment discontinuation and clinical evaluation.
* At M3, M6, M9 and M12: • Number of falls, all treatment schedule, record of major bleeding events, record of any other bleeding events, record of other serious events, record of other non-major events, treatment discontinuation, and social and medical environment.
* Only M6 and M12: Renal function (both Cockcroft-Gault, chronic Kidney Disease, epidemiology Collaboration "CKD EPI" and the four variable modification of Diet in renal Disease equation "MDRD")

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 80 years and older.
* Patients with non-valvular atrial fibrillation (documented on electrocardiography or other medical evidence like medical chart, hospital discharge note, physician's letter within 3 years before enrollment).
* Followed in geriatric settings (office consultation, acute care, rehabilitation settings and nursing homes).
* Newly treated (less than 6 months) with Apixaban (5mg twice daily (or 2.5 mg twice daily for patients with 2 of the following criteria : age > 80 years, creatinine > 133 μmol/l, weight < 60 kg)

Exclusion Criteria:

* Patient refusing to participate.
* Participation to a clinical trial.
* Contraindication to use of Apixaban as described in the Summary of Product Characteristics .

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients newly treated with Apixaban for non-valvular atrial fibrillation (no mechanical heart valves, no known moderate or severe mitral stenosis)
Sampling Method: Non-Probability Sample
Enrollment: 977 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Assessment of the incidence of bleeding events | 12 months

SECONDARY OUTCOMES:
To determine bleeding risk according (ATRIA bleeding) score | 12 months
Assessment of compliance with treatment by (Apixaban) according (Morisky) Score | 12 months
To quantifie risk of hemorrhage according (HEMORR₂HAGES) Score | 12 months
Assessment of the risk of bleeding according the (HAS-BLED) Score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD PhD, Study Chair — Geriatric Department, Broca hospital
Locations (1):
- Geriatric Department, Broca Hospital, Paris, IIe-de-France, France